CLINICAL TRIAL: NCT01098617
Title: The Effect of Antiaggregant, Anticoagulant and Nonsteroidal Antiinflammatory Therapy on Endoscopic Biliary Sphincterotomy Induced Bleeding
Brief Title: Antihemostatic Therapy and Endoscopic Biliary Sphincterotomy Induced Bleeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yuksek Ihtisas Hospital (Other)
Responsible Party: Yuksek Ihtisas Hospital, Yuksek Ihtisas Hospital Gastroenterology Department
Other Study IDs: PMS207
Record Dates: First submitted 2010-04-01; First posted 2010-04-05 (Estimated); Last update posted 2010-04-05 (Estimated); Status verified 2010-04

CONDITIONS: Endoscopic Biliary Sphincterotomy; Bleeding
Keywords: endoscopic sphincterotomy; hemorrhage; nonsteroidal antiinflammatory agents; antiaggregants; anticoagulants; Endoscopic biliary sphincterotomy induced bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- hemorrhage: The patients who had bleeding induced by endoscopic sphincterotomy

SUMMARY:
The aim of the study is to observe the effects of antihemostatic therapy including nonsteroidal antiinflammatory, anticoagulant and antiaggregant therapy and other patient and procedure related factors on the risk of endoscopic biliary sphincterotomy induced bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization
* Endoscopic sphincterotomy
* The patients whose warfarin treatment was stopped and INR was normalized prior to examination

Exclusion Criteria:

* The patients who had undergone endoscopic cholangiography with no sphincterotomy
* Outpatient procedures

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who had undergone endoscopic sphincterotomy
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Bleeding induced by endoscopic biliary sphincterotomy | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Meral Akdoğan, MD, Principal Investigator — Turkiye Yuksek Ihtisas Hospital Gastroenterology Department; Ibrahim Koral Onal, MD, Principal Investigator — Turkiye Yuksek Ihtisas Hospital Gastroenterology Department; Erkan Parlak, MD, Study Director — Turkiye Yuksek Ihtisas Hospital Gastroenterology Department
Locations (1):
- Turkiye Yuksek Ihtisas Hospital, Ankara, Turkey (Türkiye)